CLINICAL TRIAL: NCT04931966
Title: Comparision of IPACK and Periarticular Block With Adductor Block Alone After Total Knee Artroplasty: a Prospective Randomized Trial on Pain and Knee Function After Total Knee Artroplasty
Brief Title: Comparision of IPACK and Periarticular Block With Adductor Block Alone After Total Knee Artroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karaman Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 02-202l/04:
Record Dates: First submitted 2021-06-09; First posted 2021-06-18 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Osteo Arthritis Knee
Keywords: Total knee arthroplasty; Peri articular infiltration; Ipack block; Adductor canal block
MeSH Terms: interventions — Dental Occlusion

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Active Comparator): Adductor canal block
  Interventions: Procedure: block; Procedure: adductor canal block
- Group B (Active Comparator): Adductor canal block plus IPACK
  Interventions: Procedure: block; Procedure: adductor canal block; Procedure: Adductor Canal Block plus IPACK Block
- Group C (Active Comparator): Adductor canal block plus PAI
  Interventions: Procedure: block; Procedure: adductor canal block; Procedure: adductor Canal Block plus PAI Block

INTERVENTIONS:
Procedure: block — Adductor canal block
Procedure: adductor canal block — adductor canal block bupivacain
Procedure: Adductor Canal Block plus IPACK Block — Adductor Canal Block plus IPACK Block using bupivacaine
  Arms: Group B
Procedure: adductor Canal Block plus PAI Block — Adductor Canal Block plus PAI Block using bupivacaine
  Arms: Group C

SUMMARY:
105 patients ASA I-III, undergoing total knee arthroplasty under spinal anesthesia, will be randomly assigned into one of three groups, namely group A (n=35), where an adductor canal block, group B (N:35) where an adductor canal block with IPCAK, and group C (n=35) where an adductor canal block with PAI will be performed preoperatively. All patients will receive a standardized multimodal approach. NRS scores will be evaluated in static and dynamic conditions during the first 48 hours postoperatively.

DETAILED DESCRIPTION:
Total knee replacement (TKP) is accepted as one of the major orthopedic surgery that most patients suffer from pain in the postoperative period. The primary aim of this research is to compare the analgesic efficacy of infiltration between the popliteal artery and capsule of the knee(IPACK) with the periarticular block when an additional adductor canal block is used. In the literature, adductor canal block(ACB) and sciatic nerve block are used as part of multimodal analgesia for postoperative pain management of patients undergoing TKP. Nevertheless, ACB is found less effective for pain originating from the posterior part of the knee. Sciatic nerve block and periarticular injection(PAI) are commonly used blocks to improve the analgesic effect of ACB. Besides this, ACB is effective for pain originated from the posterior part of the knee. IPACK block is performed under ultrasound guidance and targets the articular branches of tibial, common peroneal, and obturator nerves with sparing lower extremity motor function.

Patients scheduled for knee surgery under spinal anesthesia are included fort his study. All groups will be applied 0.03 mg/kg midazolam iv, then spinal anesthesia will be applied to 15 mg 0.5 % heavy bupivacaine. Three groups of 105 patients will be included in the study.

Adductor Canal Block (ACB) (Group A ) (n:35): After the patients are given the supine position, under the guidance of the ultrasound linear probe, 10-15cm proximal to the knee joint, under the sartorius muscle, next to the femoral artery. After the saphenous is observed, 0.25% 20 mL of bupivacaine will be given

Adductor + İPACK Grup ( group B) (n: 35): Adductor canal 0.25% 20 mL of bupivacaine will be administered. After the knee is flexed, after the convex probe is placed in the popliteal space, 20 ml of 0.25% bupivacaine will be injected into the area between the popliteal artery and the femur called IPACK

Adductor + PAI ( group C) (n: 35): Adductor canal 0.25% 20 mL of bupivacaine will be administered. Patients will receive 60 ml of local anesthetic cocktail intraoperatively by the surgeon. At the end of the operation to the peri-articular area (posterior capsule, collateral ligament, quadriceps muscle). Cocktail consists of 40 ml 0.25% bupivacaine + 8 ml 8 mg morphine+12 ml saline.

Routine multimodal analgesia will be used for postoperative analgesia

ELIGIBILITY:
Inclusion Criteria:

* Physical status according to American Society of Anesthesiologists (ASA) I-III
* Patients scheduled for total knee arthroplasty

Exclusion Criteria:

* Previous operation on same knee
* Hepatic or renal insufficiency
* Younger than 18 years old and older than 85
* Patients undergoing general anesthesia
* Allergy or intolerance to one of the study medications
* BMI > 40
* ASA IV
* Chronic gabapentin/pregabalin use (regular use for longer than 3 months)
* Chronic opioid use (taking opioids for longer than 3 months, or daily oral morphine equivalent of >5mg/day for one month)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2021-08-08 (Actual); Study Completion 2021-08-17 (Actual)

PRIMARY OUTCOMES:
NRS scores | 48 hours
  Numerical Rating Scale (NRS) scores (Range 0-10, 0=no pain, 10=the worse pain ever)

SECONDARY OUTCOMES:
Opioid consumption | 4-6-8-12-24 and 48 hours
  Analgesic consumption at 4-6-8-12-24 and 48 hours
Range of knee motion | 48 hours
  Degrees of flexion
Complications | 48 hours
  Complications
Patient satisfaction | 48 hours
  Patients asked whether they would choose the same anaesthetic management in a future operation: Yes/No
Incidence of adverse events related to nerve block procedures | Post-op 24 to 72 hours
  muscle weakness, systemic toxicity
Rate of postoperative nausea and vomiting | Post-op 24 to 48 hours
  nausea, vomiting
Patient mobilization | 2 days
  Patient reporting time of first standing to the side of the bed and time up and go test 2 days

CONTACTS AND LOCATIONS:
Locations (1):
- Karaman Training and Research Hospital, Karaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kertkiatkachorn W, Kampitak W, Tanavalee A, Ngarmukos S. Adductor Canal Block Combined With iPACK (Interspace Between the Popliteal Artery and the Capsule of the Posterior Knee) Block vs Periarticular Injection for Analgesia After Total Knee Arthroplasty: A Randomized Noninferiority Trial. J Arthroplasty. 2021 Jan;36(1):122-129.e1. doi: 10.1016/j.arth.2020.06.086. Epub 2020 Jul 2. PMID 32694032
- [Background] Kim DH, Beathe JC, Lin Y, YaDeau JT, Maalouf DB, Goytizolo E, Garnett C, Ranawat AS, Su EP, Mayman DJ, Memtsoudis SG. Addition of Infiltration Between the Popliteal Artery and the Capsule of the Posterior Knee and Adductor Canal Block to Periarticular Injection Enhances Postoperative Pain Control in Total Knee Arthroplasty: A Randomized Controlled Trial. Anesth Analg. 2019 Aug;129(2):526-535. doi: 10.1213/ANE.0000000000003794. PMID 30234517